CLINICAL TRIAL: NCT00814632
Title: A Clinical Trial Of CC-10004 For The Treatment Of Vulvodynia
Brief Title: CC-10004 For The Treatment Of Vulvodynia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kenneth Peters, MD (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor-Investigator, Kenneth Peters, MD, Principal Investigator, Corewell Health East
Organization: Corewell Health East (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-134
Record Dates: First submitted 2008-12-23; First posted 2008-12-25 (Estimated); Results first posted 2014-09-29 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Vulvodynia
Keywords: vulvodynia; pelvic pain; vulvar pain
MeSH Terms: conditions — Vulvodynia; Pelvic Pain | interventions — apremilast; Drug Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study Drug CC 10004 (Experimental): Study drug CC-10004 20mg taken orally twice a day.
  Interventions: Drug: CC-10004

INTERVENTIONS:
Drug: CC-10004 — CC-10004 20 mg. twice a day for 12 weeks
  Other Names: Study Drug

SUMMARY:
Vulvodynia is characterized by persistent vulvar pain, which often occurs upon touch or pressure. The cause of vulvodynia is unknown but is presumed to involve many factors. Some of these factors may include altered immune response, infections, altered vaginal acid-base balance, allergic reactions and psychosexual disorders. Women are generally treated with medications such as anti-histamines, anti-depressants and anti-inflammatories, or with physical therapy to minimize symptoms. Other therapies for vulvodynia include topical agents (lidocaine, or compounded medications such as baclofen, gabapentin and amitriptyline), oral medications (gabapentin, pregabalin, calcium citrate), complementary therapies (yoga, guided imagery, cognitive behavioral therapy) or a low-oxalate diet, but these are often ineffective. Surgery for vulvodynia may be helpful in the hard to manage cases, but is utilized as a last resort.

DETAILED DESCRIPTION:
CC-10004 is a well-tolerated, selective PDE4 inhibitor with a demonstrated inhibitory effect on inflammatory mediators and is under development for the treatment of inflammatory and immune mediated conditions.

This is an open-label, one arm, phase II study at William Beaumont Hospital. Twenty female subjects aged 18 or older meeting criteria for diagnosis of vulvodynia or vulvar vestibulitis (vestibulodynia) will be treated with CC-10004 at 20mg orally twice a day for 12 weeks.The patient will be seen for a total of ten visits by the study coordinator.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must understand and voluntarily sign and date the appropriate Informed Consent document.
2. Female who is ≥ 18 years of age and <70 years of age.
3. Participant must be able to adhere to the study visit schedule and other protocol requirements.
4. Participant must have vulvodynia--vulvar pain at 2 or more sites tested of at least 3 or greater on a 0-10 Likert scale.
5. Subject -reported vulvar pain for at least 3 months prior to enrollment.
6. Participant who is currently taking narcotics for pelvic pain must be on a stable regimen for 3 months prior to enrollment in the study.
7. Females of childbearing potential (FCBP) must have a negative urine pregnancy test at screening/baseline (Visit 1). In addition, sexually active FCBP must agree to use TWO of the following adequate forms of contraception while on study medication: oral, injectable, or implantable hormonal contraceptives; tubal ligation; intrauterine device; barrier contraceptive with spermicide; or vasectomized partner. A FCBP must agree to have pregnancy tests every 28 days while on study medication.
8. Subject must meet the following laboratory criteria:

   * Hemoglobin > 9 g/dL
   * Hematocrit ≥ 27%
   * White blood cell (WBC) count ≥ 3000 /mL (≥ 3.0 X 109/L) and < 20,000/mL (< 20 X 109/L)
   * Neutrophils ≥ 1500 /mL (≥ 1.5 X 109/L)
   * Platelets ≥ 100,000 /mL (≥ 100 X 109/L)
   * Serum creatinine ≤ 1.5 mg/dL (≤ 132.6 μmol/L)
   * Total bilirubin £ 2.0 mg/dL
   * Aspartate transaminase (AST [serum glutamic oxaloacetic transaminase, SGOT]) and alanine transaminase (ALT [serum glutamate pyruvic transaminase, SGPT]) < 1.5x upper limit of normal (ULN)

Exclusion Criteria:

1. Pregnant or lactating females
2. History of any clinically significant cardiac, endocrinologic, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic conditions, or other major diseases
3. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
4. History of active Mycobacterium tuberculosis infection (any subspecies) within 3 years prior to the screening visit. Infections that occurred > 3 years prior to entry must have been effectively treated.
5. Positive TB skin test (Mantoux test)
6. History of incompletely treated latent Mycobacterium tuberculosis infection as indicated by a positive positive Purified Protein Derivative [PPD] skin test or in vitro test [T-SPOT®. TB, QuantiFERON Gold®] or chest x-ray.
7. Clinically significant abnormality on the chest x-ray (CXR) at screening.
8. Use of any investigational medication within 28 days prior to randomization or 5 half-lives if known (whichever is longer)
9. Any clinically significant abnormality on 12-lead ECG at screening
10. Positive human immunodeficiency virus (HIV), hepatitis B, or hepatitis C laboratory test result indicating active infection at screening.
11. History of malignancy within previous 5 years (except for treated basal-cell skin carcinoma(s) and/or fewer than 3 treated squamous-cell skin carcinomas)
12. History of a vestibulectomy

Ages: 18 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-12; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth M Peters, M.D., Principal Investigator — Beaumont Hospitals
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Drug CC 10004: Study drug CC-10004 20mg taken orally twice a day for 12 weeks.
Period: Overall Study
Arm/Group | Study Drug CC 10004
Started | 9 (Ten were allocated to treatment intervention however one was not treated due to lactose allergy.)
Completed | 7 (Two subjects withdrew early due to lack of efficacy.)
Not Completed | 2
Not completed — Lack of Efficacy | 2

BASELINE CHARACTERISTICS:
Arm/Group | Study Drug CC 10004
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Global Response Assessment
Description: The primary efficacy measure was a Global Response Assessment (GRA), a subject completed questionnaire that measures improvement in overall symptoms. The GRA is a 7-point scale the allows the subject to respond to the question: "As compared to when you started the study, overall how do you feel? The responses are: Markedly Improved - 7, Moderately Improved - 6, Mildly Improved - 5, Same - 4, Mildly Worse - 3, Moderately Worse - 2, Markedly Worse - 1.
  The primary outcome showing response to treatment was the number of subjects that were moderately or markedly improved on the GRA scale.
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Study Drug CC 10004
Number analyzed (Participants) | 7
participants | 5

ADVERSE EVENTS:
Arm/Group | Study Drug CC 10004
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

LIMITATIONS AND CAVEATS:
Small pilot study without placebo arm. Only 7 subjects completed treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes